CLINICAL TRIAL: NCT01247181
Title: Improving Adherence to HAART Using Mobile Phone Text Messages
Brief Title: Cameroon Mobile Phone SMS Trial
Acronym: CAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Lawrence Mbuagbaw, MD, MPH, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CAMPS; PACTR201011000261458 (Registry Identifier: Pan-African Clinical Trials Registry)
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Adherence; HIV
Keywords: compliance; observance; mobile phone; SMS; text message; ARV; HAART; AIDS
MeSH Terms: conditions — Patient Compliance; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile phone text message (Experimental)
  Interventions: Other: Mobile phone text message
- No Mobile phone text message (Active Comparator): Usual care provided at clinic
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Mobile phone text message — Weekly message with motivational content
  Other Names: SMS; Texto; Text message
  Arms: Mobile phone text message
Other: Usual care — Usual care provided at clinic
  Other Names: Routine care
  Arms: No Mobile phone text message

SUMMARY:
The investigators hypothesize that sending weekly motivational text messages to people infected with HIV will encourage them to take their medication, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* On HAART for at least 1 month
* 21 years or more
* Owns a mobile phone
* Can read text messages

Exclusion Criteria:

* On HAART for less than 1 month
* Aged less than 21 years

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Adherence | Change from baseline at 6 months
  Measured using the Visual Analogue Scale, Self Report and Pharmacy Refill Data

SECONDARY OUTCOMES:
Weight | Change from baseline at 6 months
Body Mass Index | Change from baseline at 6 months
CDC classification | Change from baseline at 6 months
WHO Classification | Change from baseline at 6 months
Mortality | 6 months
  All cause mortality
CD4 count | Change from baseline at 6 months
Viral load | Change from baseline at 6 months
Quality of life | Change from baseline at 6 months
  Measured using the SF-12 quality of life form

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mbuagbaw, MD, MPH, Principal Investigator — Centre for the Development of Best Practices in Health; Pierre Ongolo-Zogo, MD, BSc, Study Director — Centre for the Development of Best Practices in Health
Locations (1):
- Yaounde Central Hospital Accredited Treatment Centre, Yaoundé, Centre Region, Cameroon

REFERENCES:
- [Derived] Mbuagbaw L, Thabane L, Ongolo-Zogo P, Lester RT, Mills EJ, Smieja M, Dolovich L, Kouanfack C. The Cameroon Mobile Phone SMS (CAMPS) trial: a randomized trial of text messaging versus usual care for adherence to antiretroviral therapy. PLoS One. 2012;7(12):e46909. doi: 10.1371/journal.pone.0046909. Epub 2012 Dec 6. PMID 23236345
- [Derived] Mbuagbaw L, Thabane L, Ongolo-Zogo P, Lester RT, Mills E, Volmink J, Yondo D, Essi MJ, Bonono-Momnougui RC, Mba R, Ndongo JS, Nkoa FC, Ondoa HA. The Cameroon mobile phone SMS (CAMPS) trial: a protocol for a randomized controlled trial of mobile phone text messaging versus usual care for improving adherence to highly active anti-retroviral therapy. Trials. 2011 Jan 7;12:5. doi: 10.1186/1745-6215-12-5. PMID 21211064